CLINICAL TRIAL: NCT00272103
Title: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled Dose Finding Study in 4 Parallel Groups to Establish the Efficacy and Safety of an Eight Week Treatment With Itopride Three Times Daily Compared to Placebo in Patients Suffering From Functional Dyspepsia
Brief Title: Itopride in Functional Dyspepsia:a Dose Finding Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Adelaide Hospital (Other)
Collaborators: Knoll Pharmaceuticals, Germany (now Abbott) (Unknown); University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KD20003
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2005-11

CONDITIONS: Functional Dyspepsia
Keywords: functional dyspepsia; non ulcer dyspepsia; drug treatment
MeSH Terms: interventions — itopride; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Itopride (drug)

SUMMARY:
This study aims to determine the efficacy and optimal dose of the prokinetic itopride for the treatment of patients with functional dyspepsia.

The study will test in patients with functional dyspepsia the hypothesis that itopride is superior to placebo with regard to the improvement of symptoms.

DETAILED DESCRIPTION:
Treatment of patients with functional dyspepsia remains unsatisfactory. We will assess the efficacy of Itopride, a D2 antagonist with acetylcholinesterase effects in patients with functional dyspepsia.

Patients with functional dyspepsia will be randomized to Itopride (50, 100 or 200 mg tid) or placebo. After 8 weeks of treatment, three primary efficacy endpoints will be analyzed: a) change of the severity of functional dyspepsia symptoms (assessed by the Leeds Dyspepsia Questionnaire), b) patient's global assessment of efficacy (proportion of patients symptom-free or markedly improved)and c) improvement of pain and/or fullness by at least one grade on a 5-grade scale.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of functional dyspepsia (Rome criteria) -

Exclusion Criteria:

structural or biochemical abnormalities explaining the symptoms, concomitant symptoms of gastroesophageal reflux disease or irritable bowel syndrome dominating the clinical picture

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2000-12; Study Completion 2002-01

PRIMARY OUTCOMES:
After 8 weeks of treatment:
Change of the severity of functional dyspepsia symptoms assessed by the Leeds Dyspepsia Questionnaire)
Patient's global assessment of efficacy (proportion of patients symptom-free or markedly improved)
Improvement of pain and/or fullness by at least one grade on a 5-grade scale.

SECONDARY OUTCOMES:
Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Gerald J Holtmann, MD, Principal Investigator — Royal Adelaide Hospital, University of Adelaide
Locations (1):
- University Hospital Essen, Essen, Hesse, Germany

REFERENCES:
- [Result] Holtmann G, Talley NJ, Liebregts T, Adam B, Parow C. A placebo-controlled trial of itopride in functional dyspepsia. N Engl J Med. 2006 Feb 23;354(8):832-40. doi: 10.1056/NEJMoa052639. PMID 16495395